CLINICAL TRIAL: NCT00400478
Title: A Multicentre, Randomized Phase III Study of Rituximab as Maintenance Treatment Versus Observation Alone in Patients With Aggressive B-cell Lymphoma: NHL-13
Brief Title: A Multicentre, Randomized Phase III Study of Rituximab as Maintenance Treatment Versus Observation in Patients With Aggressive B-cell Lymphoma: NHL-13
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHL-13 (ML18223)
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Diffuse Large B-Cell Lymphoma (DLBCL); Follicular NHL Grade 3b
Keywords: DLBCL; NHL 13; Rituximab; maintenance
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Treatment
  Interventions: Drug: Rituximab
- B (No Intervention): Observation

INTERVENTIONS:
Drug: Rituximab — Rituximab 375mg/m2 i every 8 weeks for two years (12 infusions)
  Arms: A

SUMMARY:
This is a randomized, open label, phase III study to evaluate the ability of rituximab maintenance therapy to prolong event-free survival in aggressive NHL.

Patients will be screened after successful standard induction therapy (CR or Cru following standard R-CHOP-like therapy with 8 infusions of rituximab plus CHOP-like chemotherapy (4-8 cycles). Patients will be followed until an event occurs as defined in the protocol. To evaluate the clinical efficacy of rituximab maintenance therapy as compared to observation in patients with aggressive B-cell Non-Hodgkins lymphoma or follicular lymphoma grade 3b who have achieved a complete remission after appropriate first-line therapy, measured by event-free survival (EFS), 440 patients with DLCBL or follicular NHL grade 3 (220 per arm) will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* 4 to 8 cycles R-CHOP/like, total of 8x Rituximab
* CR, CRu
* ECOG/ 0.1 or 2
* Known IPI at time of diagnosis
* Age > 18 years
* Negative pregnancy test
* Men must agree not to father a child during the therapy

Exclusion Criteria:

* Transformed lymphoma
* Secondary malignancy
* Evidence of CNS - involvement
* Significant cardiac disease
* Creatinine > 2.0 mg/dl
* HIV, Hepatitis positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2006-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
event free survival | 4 years

SECONDARY OUTCOMES:
progression free survival, overall survival and safety | four years

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Jaeger, Prof. Dr., Principal Investigator — Medical University of Vienna
Locations (130):
- Australia (5):
  - Border Medical Oncology, Wodonga, Victoria
  - Concord Repatriation General Hospital, Concord
  - Gosford Hospital, Gosford
  - Greenslopes Hospital, Greenslopes
  - Prince of Wales Hospital, Sydney
- Austria (36):
  - Krankenhaus Oberpullendorf, Oberpullendorf, Burgenland
  - Krankenhaus Oberwart, Oberwart, Burgenland
  - A.ö. Krankenhaus der Landeshauptstadt St. Pölten, Sankt Pölten, Lower Austria
  - A.ö. Krankenhaus der Statutarstadt Wr. Neustadt, Wiener Neustadt, Lower Austria
  - St. Johanns LK, Salzburg, Salzburg
  - A.ö. Landeskrankenhaus Steyr, Steyr, Styria
  - Bezirkskrankenhaus Kufstein, Endach, Tyrol
  - A.oe.Bezirkskrankenhaus Hall, Hall in Tirol, Tyrol
  - Universitätsklinik Innsbruck/ Klinik für Innere Medizin, Innsbruck, Tyrol
  - Krankenhaus d. Barmherzigen Schwestern Linz, Linz, Upper Austria
  - Krankenhaus der Elisabethinen Linz, Linz, Upper Austria
  - KH Barmherzige Schwestern Ried, Ried, Upper Austria
  - Klinikum Kreuzschwestern Wels GmbH, Wels, Upper Austria
  - KH Barmherzige Brüder, Vienna, Vienna
  - Krankenhaus der Stadt Wien Rudolfsstiftung, Vienna, Vienna
  - AKH Wien / Hämatologie u. Hämostaseologie, Vienna, Vienna
  - Kaiser-Franz-Josef-Spital, Vienna, Vienna
  - Krankenhaus der Stadt Wien Lainz, Vienna, Vienna
  - Hanusch-Krankenhaus, Vienna, Vienna
  - Wilhelminenspital, Vienna, Vienna
  - Sozialmedizinisches Zentrum Ost - Donauspital, Vienna, Vienna
  - Landeskrankenhaus Feldkirch, Feldkirch, Vorarlberg
  - LKH Bregenz, Bregenz
  - KH Dornbirn, Dornbirn
  - A.ö. Landeskrankenhaus Fürstenfeld, Fürstenfeld
  - Universitätsklinikum Graz, Graz
  - LKH Hohenems, Hohenems
  - Universitaetsklinik Innsbruck, Innsbruck
  - Landeskrankenhaus Klagenfurt, Klagenfurt
  - A.ö. Landeskrankenhaus Leoben, Leoben
  - Krankenhaus der Stadt Linz, Linz
  - LKH Weinviertel Mistelbach, Mistelbach
  - LKH Villach, Villach
  - LKH Vöcklabruck, Vöcklabruck
  - KH Waidhofen/Thaya, Waidhofen an der Thaya
  - BKH Zams, Zams
- Bosnia and Herzegovina (2):
  - Clinical Centre University Sarajevo, Sarajevo
  - University Center Tuzla, Tuzla
- Brazil (4):
  - Centro Goiano de Oncologia, Goiânia
  - Hospital Santa Izabel, Salvador
  - Hospital das Clinicas FMUSP, São Paulo
  - Hospital deas Clinical FMUSP, São Paulo
- Bulgaria (3):
  - UMHAT "St. George" Plodviv, Plovdiv
  - Nat. Centre of Hematology and Transfusiology Sofia, Sofia
  - MHAT "St. Marina" Varna, Varna
- China (6):
  - Chinese PLA General hospital, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - Harbin Institue, Harbin
  - Jiangsu Cancer Hospital, Nanjing
  - Changhai Hospital, Shanghai
  - Shanghai Ruijin Hospital, Shanghai
- Croatia (3):
  - Clinical Hopital Center Zagreb, Zagreb
  - Clinical Hospital Dubrava, Zagreb
  - Clinicall Hospital "Merkur", Zagreb
- Czechia (11):
  - Nemocnice Boskovice s.r.o., Boskovice
  - Faculty Hospital Brno, Brno
  - Univ. Hospital and Med. School Hradec Kralove, Kralove
  - Onkologické Centrum J.G. Mendela, Novi Jicin
  - Fakultni Nemocnice Olomouc, Olomouc
  - Hospital Opava, Opava
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Charles University Hospital, Prague
  - Faculty Hospital Binohrady FNKV, Prague
  - University Hospital Motol, Prague
  - RTO MN Usti n. Labem, Ústí nad Labem
- Estonia (2):
  - North Estonian Regional Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- Israel (4):
  - Soroka Medical Centre, Beersheba
  - Rambam Medical Centre, Haifa
  - Rabin Medical Centre, Petah Tikva
  - Kaplan Medical Centre, Rehovot
- Riga Hematology Center, Riga, Latvia
- Malaysia (2):
  - Hospital Ampang, Ampang
  - Hospital University Kebangsaan Malaysia, Kuala Lumpur
- Mexico (6):
  - ISSSTE Hospital Regional de Leon, León
  - Hospital Espanol de Mexico, Mexico City
  - Hospital General de Mexico, Mexico City
  - Instituto National de Cancerologia, Mexico City
  - Hospital Regional Monterrey, ISSTE, Monterrey
  - ISSSTEP Puebla, Puebla City
- Clinical Centre Skopje, Skopje, North Macedonia
- Peru (2):
  - Hospital Carlso alberto seguin escobedo Arequipa, Arequipa
  - Hospital Alberto Sabogal sooguren Callao, Callao
- Romania (4):
  - Coltea Hospital, Bucharest
  - University Emergency Center Bucharest, Bucharest
  - Clinic Judatean de Urgenta Brasov, Târgu Mureş
  - Emergency County Clinical Hospital, Târgu Mureş
- Russia (7):
  - Belgorod regional Clinical Hospital, Belgorod
  - Moscow Regional Clinical Research Institute, Moscow
  - Botkin City Clinical Hospital, Moscow
  - Leningrad regional Cliniacal Hospital, Saint Petersburg
  - SPB Pavlov State Medical University, Saint Petersburg
  - Republican Clinic Oncology Dispensary, Ufa
  - Novgorod Regional Clinical Hospital, Veliky Novgorod
- Serbia (4):
  - Clinical centre of Serbia, Belgrade, Belgrade
  - Institute of Oncology Sremska Kamenica, Kamenitz
  - Clinical Centre Nis, Niš
  - Clinical Centre Novi Sad, Novisad
- Slovakia (4):
  - National Cancer Institut Bratislava, Bratislava
  - OUSA Bratislava, Bratislava
  - Východoslovenský onkolgický ústav, Košice
  - Martinská fakultná nemocnima, Martin
- Institut of Oncology Ljubljana, Ljubljana, Slovenia
- South Africa (2):
  - Hopelands Cancer Centre, Pietremarizburg
  - Wilgers Oncology Centre, Pretoria
- Sweden (4):
  - Falun Hospital, Falun
  - Sunderby Hospital, Luleå
  - Sundsvall Hospital, Sundsvall
  - Uddevalla Hospital, Uddevalla
- Taiwan (3):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
  - Taichung Veterans General Hospital, Taipei
- Thailand (7):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao College of Medicine, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriray Hospital, Bangkok
  - Chiang Mai University, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Songklanagrarind Hospital, Songkhla
- Turkey (Türkiye) (4):
  - Ankara University, School of Medicine, Ankara
  - Osmangazi Univ. school of Medicine, Eskişehir
  - Gaziantep University School of Medicine, Gaziantep
  - Ericyes Univ. Med. School, Kayseri

REFERENCES:
- [Result] Jaeger U, Trneny M, Melzer H, Praxmarer M, Nawarawong W, Ben Yehuda D, Goldstein D, Mihaljevic B, Ilhan O, Ballova V, Hedenus M, Hsiao LT, Au WY, Burgstaller S, Weidinger G, Keil F, Dittrich C, Skrabs C, Klingler A, Chott A, Fridrik MA, Greil R; AGMT-NHL13 Investigators. Rituximab maintenance for patients with aggressive B-cell lymphoma in first remission: results of the randomized NHL13 trial. Haematologica. 2015 Jul;100(7):955-63. doi: 10.3324/haematol.2015.125344. Epub 2015 Apr 24. PMID 25911553
- [Result] Jaeger U, Praxmarer M, Greil R; AGMT-NHL13 investigators. Response to comment by P. Vassilakopoulos and colleagues. Haematologica. 2015 Nov;100(11):e482. doi: 10.3324/haematol.2015.134288. No abstract available. PMID 26521299
- See also: AGMT — http://www.agmt.at
- Available data/document: Clinical Study Report — https://www.clinicaltrialsregister.eu/ctr-search/search;jsessionid=cJHnlkSBP30JjfQV2K-KXCK3mdjOE64o0FAsUcmzHmslzlaX5yhQ!675812678